CLINICAL TRIAL: NCT03902392
Title: Oral Human Administration of Red Grape Polyphenol in Nickel-mediated Allergic Contact Dermatitis: an in Vitro Study
Brief Title: Red Grape Polyphenol Oral Administration to Women Affected by Nickel-mediated Allergic Contact Dermatitis
Acronym: Grapolyphen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bari (Other)
Responsible Party: Principal Investigator, Thea Magrone, Aggregate Professor of Immunology, University of Bari
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 5480
Record Dates: First submitted 2019-02-14; First posted 2019-04-04 (Actual); Results first posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Allergic Contact Dermatitis
Keywords: Allergic contact dermatitis; Cytokines; Cellular and molecular rehabilitation; Immune response; Nickel; Polyphenols
MeSH Terms: conditions — Dermatitis, Allergic Contact

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NATUR-OX Group (A) (Active Comparator): Administration, for three months (T1), of NATUR-OX® capsule/day. NATUR-OX® which is a dietary supplement containing grape seed extracts from Nero di Troia (Vitis vinifera). Each capsule contains 280 mg of proanthocyanidins where Ni contamination of capsule is below 0.24 ppm
  Interventions: Dietary Supplement: NaturOx Group (A)
- Placebo Group (B) (Placebo Comparator): Administration with placebo one capsule/daily for three months. The placebo capsules had the same appearance and composition of the supplement except for the active ingredient (polyphenols)
  Interventions: Other: Placebo Group (B)

INTERVENTIONS:
Dietary Supplement: NaturOx Group (A) — Comparison between dietary supplement and placebo
  Arms: NATUR-OX Group (A)
Other: Placebo Group (B) — Comparison between dietary supplement and placebo
  Arms: Placebo Group (B)

SUMMARY:
Nickel (Ni)-mediated allergic contact dermatitis (ACD) is a very common disease worldwide. Our previous findings demonstrated that in vitro supplementation of polyphenols, extracted from seeds of red grape (Nero di Troia cultivar), to peripheral lymphomonocytes from Ni-mediated ACD patients could reduce release of T helper (h)1 [interferon (IFN)-] and Th2 [interleukin (IL)-4] cytokines, on the one hand. On the other hand, IL-10 (an anti-inflammatory cytokine) levels increased with a reduction of IL-17 (an inflammatory cytokine). Also levels of nitric oxide (NO) decreased in response to polyphenol pretreatment.

DETAILED DESCRIPTION:
Nickel (Ni) is a transitional metal largely distributed in the environment whose continuous exposure is able to provoke local and systemic allergic contact dermatitis (ACD). Ni-mediated ACD is characterized by loss of epidermal integrity, urticaria/angioedema, flares, and itching, whose extent depends on many variables such as genetic, time of sensitization and environmental exposure.The aim of the present research is to verify whether the oral administration of polyphenols (NATUR-OX®) to patients with Ni-mediated ACD is able to modify immune parameters.

ELIGIBILITY:
Inclusion Criteria:

* Female patient; Age: 25-60 Years; Ni-mediated ACD (positive reaction to the nickel patch test)

Exclusion Criteria:

* Absence of other pathologies such as immune-mediated diseases, metabolic diseases (diabetes and obesity)
* infectious episodes in the last month and intake of immunosuppressive drugs or drugs influencing the immune response.

Ages: 25 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2018-09-10 (Actual); Study Completion 2018-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caterina CF Foti, MD, Principal Investigator — University of Bari
Locations (1):
- Thea Magrone, Bari, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Magrone T, Romita P, Verni P, Salvatore R, Spagnoletta A, Magrone M, Russo MA, Jirillo E, Foti C. In vitro Effects of Polyphenols on the Peripheral Immune Responses in Nickel-sensitized Patients. Endocr Metab Immune Disord Drug Targets. 2017 Nov 16;17(4):324-331. doi: 10.2174/1871530317666171003161314. PMID 28982342
- [Result] Johansen JD, Aalto-Korte K, Agner T, Andersen KE, Bircher A, Bruze M, Cannavo A, Gimenez-Arnau A, Goncalo M, Goossens A, John SM, Liden C, Lindberg M, Mahler V, Matura M, Rustemeyer T, Serup J, Spiewak R, Thyssen JP, Vigan M, White IR, Wilkinson M, Uter W. European Society of Contact Dermatitis guideline for diagnostic patch testing - recommendations on best practice. Contact Dermatitis. 2015 Oct;73(4):195-221. doi: 10.1111/cod.12432. Epub 2015 Jul 14. PMID 26179009
- [Result] Summer B, Stander S, Thomas P. Cytokine patterns in vitro, in particular IL-5/IL-8 ratio, to detect patients with nickel contact allergy. J Eur Acad Dermatol Venereol. 2018 Sep;32(9):1542-1548. doi: 10.1111/jdv.14931. Epub 2018 Mar 26. PMID 29524267

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NATUR-OX Group (A) | Placebo Group (B)
Started | 25 | 25
Completed | 18 | 18
Not Completed | 7 | 7
Not completed — Lost to Follow-up | 7 | 7

BASELINE CHARACTERISTICS:
Population: 7 dropouts for each group.
Groups:
- Total: Total of all reporting groups
Arm/Group | NATUR-OX Group (A) | Placebo Group (B) | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Categorical [Count of Participants; unit: Participants] — Eighteen patients received NATUR-OX (age range 28-59). Eighteen patients received placebo (age range 25-60).
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 18 | 18 | 36
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 43.7 [28 to 59] | 42.5 [25 to 60] | 42.5 [25 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 36
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 18 | 18 | 36
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants] — Number of patients enrolled who are Italian.
  Participants
    Italy | 18 | 18 | 36
Evaluation of IFN-γ at T0 [Mean (Standard Deviation); unit: pg/ml] — Twenty-five patients were enrolled, and they were administered with polyphenols (NATUR-OX (A), instead other 25 patients were enrolled to assume placebo (B). From each group 7 dropouts occurred.
  pg/ml | 14.53 (3.85) | 16.03 (3.521) | 15.28 (3.72)
Evaluation of IL-17 at T0 [Mean (Standard Deviation); unit: pg/ml] | 97.58 (5.576) | 95.34 (3.982) | 96.46 (4.91)
Evaluation of IL-4 at T0 [Mean (Standard Deviation); unit: pg/ml] | 109.1 (8.944) | 110.7 (8.805) | 109.87 (8.78)
Evaluation of IL-10 at T0 [Mean (Standard Deviation); unit: pg/ml] | 14.19 (3.494) | 15.86 (3.847) | 15.03 (3.72)
Evaluation of PTX3 at T0 [Mean (Standard Deviation); unit: pg/ml] | 410.7 (46.34) | 415.6 (52.73) | 413.11 (48.98)
Evaluation of No concentrations at T0 [Mean (Standard Deviation); unit: pg/ml] | 2.401 (1.140) | 2.380 (1.233) | 2.39 (1.17)

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of Serum Biomarker Concentrations at the Time of Enrollment (T0)
Description: At the time of enrollment (T0) concentrations of serum biomarkers (pg/ml) (IFN-γ, IL-17, IL-4, IL-10, PTX3 and NO) will be evaluated in patients of which, one group (A) will assume polyphenols (NATUR-OX ) while the other group (B) will assume placebo. Of note, from each group 7 spontaneously dropouts occurred. An ELISA method will be use to analyze and to assess serum biomarker concentrations.
Time Frame: Baseline (T0)
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | NATUR-OX Group (A) | Placebo Group (B)
Number analyzed (Participants) | 18 | 18
pg/ml
  IFN-γ (measurement unit: pg/ml) | 14.53 (3.85) | 16.03 (3.521)
  IL-4 (measurement unit: pg/ml) | 109.1 (8.944) | 110.7 (8.805)
  IL-17(measurement unit: pg/ml) | 97.58 (5.576) | 95.34 (3.982)
  IL-10 (measurement unit: pg/ml) | 14.19 (3.494) | 15.86 (3.847)
  PTX3 (measurement unit: pg/ml) | 410.7 (46.34) | 415.6 (52.73)
  NO concentration (measurement unit: pg/ml) | 2.401 (1.140) | 2.380 (1.233)

2. Secondary Outcome: Evaluation of Serum Biomarker Concentrations at the End of the Treatment (T1)
Description: Serum biomarkers (IFN-γ, IL-17, IL-4, IL-10, PTX3 and NO) (pg/ml) in the same patients of both groups A and B whose received for 3 months Polyphenols (NATUR-OX) and placebo, respectively, were evaluated. To analyze serum biomarkers an ELISA method were used .
Time Frame: After 3 months (T1)
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | NATUR-OX Group (A) | Placebo Group (B)
Number analyzed (Participants) | 18 | 18
pg/ml
  IFN-γ (measurement unit: pg/ml) | 10.41 (3.964) | 17.29 (3.687)
  IL-4 (measurement unit: pg/ml) | 79.57 (8.770) | 112.2 (8.840)
  IL-17 (measurement unit: pg/ml) | 51.36 (5.374) | 100.6 (4.519)
  IL-10 (measurement unit: pg/ml) | 25.67 (5.586) | 11.19 (2.737)
  PTX3 (measurement unit: pg/ml) | 365.3 (46.08) | 455.9 (50.05)
  NO concentration (measurement unit: pg/ml) | 1.381 (0.7823) | 2.619 (1.262)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | NATUR-OX Group (A) | Placebo Group (B)
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-10-31): https://cdn.clinicaltrials.gov/large-docs/92/NCT03902392/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-31): https://cdn.clinicaltrials.gov/large-docs/92/NCT03902392/SAP_001.pdf